CLINICAL TRIAL: NCT07073092
Title: Propolis for Management of Chemotherapy-Induced Oral Mucositis in Pediatric Patients: A Randomized Controlled Clinical Trial With Biochemical Analysis
Brief Title: Propolis for Management of Chemotherapy-Induced Oral Mucositis in Pediatric Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Borham Abdelhafez Abdellatif Elkhouly, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FDASU-Rec IR/D052520
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Oral Mucositis Due to Chemotherapy
MeSH Terms: interventions — Propolis; Antifungal Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): propolis medicated jelly candy+ standard oral care (chlorohexidine and topical anti-fungal) three times daily for 21 days
  Interventions: Drug: propolis; Drug: chlorohexidine mouthwash and topical antifungal
- control group (Active Comparator): Standard oral care (chlorohexidine mouth wash and topical anti-fungal) three times daily for 21 days
  Interventions: Drug: chlorohexidine mouthwash and topical antifungal

INTERVENTIONS:
Drug: propolis — propolis medicated jelly candy.
  Arms: study group
Drug: chlorohexidine mouthwash and topical antifungal — chlorohexidine mouthwash and topical antifungal

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of propolis in the prevention of oral mucositis and reducing pain score in children undergoing chemotherapy, and assessing its impact on body mass index, pediatric quality of life and total antioxidant assay. The main question it aims to answer is:

What is the effect of propolis on oral mucositis scores in children undergoing chemotherapy?

Participants will:

Take propolis 3 times daily for 21 days follow up weekly for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Children of both genders less than 18 years receiving intensive chemotherapy.
* Oncology patients receiving intensified chemotherapy at Oncology unit, Children's Hospital, Ain Shams University, Egypt, who meet the following criteria:

  * Taking intensified chemotherapy
  * A healthy oral mucosa.

Exclusion Criteria:

* Allergy to bee products.
* Severe systemic illness unrelated to cancer (Diabetes, Hypertension, …)
* Inability to take oral medication or unwillingness to participate in the study
* Radiotherapy in the head and neck area.
* Malignant or potentially malignant lesions of the oral cavity.
* Undergoing any other procedures to prevent oral mucositis except standard oral care.
* Patients are unable to commit to the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
oral mucositis score (WHO) | 3 weeks
  Assess the effectiveness of propolis in treatment of chemotherapy induced oral mucositis in pediatric cancer patients using the WHO Scale (WHO), scoring from 0 to 4.

SECONDARY OUTCOMES:
pain (VAS) | 3 weeks
  Assess the effectiveness of propolis on pain levels. Pain will be assessed by (visual analogue scale). The P-VAS evaluation ranges from 0 to 10, where 0 indicates "no pain" and 10 indicates "the most severe pain"
body mass index | 3 weeks
  Assess the effectiveness of propolis on BMI in pediatric patients undergoing chemotherapy. Body mass index (BMI, kg/m2) was defined as the body mass (kg) divided by the square of the body height (m).
Pediatric Quality of Life | 3 weeks
  Assess the effectiveness of propolis on Pediatric Quality of Life using the Arabic validated version of Peds QL™ Inventory both Child Self Report and Parent Proxy Report.
  0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Often, 4 = Almost Always
  Scoring Method:
  1. Reverse Scoring System: 0 = 100 points, 1 = 75 points, 2 = 50 points, 3 = 25 points, 4 = 0 points 2. Domain Score Calculation: Sum all question scores within a domain and divide by the number of questions in that domain.
  3. Total PedsQL Score Calculation: Sum all domain scores and divide by the total number of questions. Higher scores indicate better quality of life.
Total anti-oxidant assay | 3 weeks
  Assess the effectiveness of propolis on total antioxidant assay in pediatric patients undergoing chemotherapy using biochemical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Docimo R, Anastasio MD, Bensi C. Chemotherapy-induced oral mucositis in children and adolescents: a systematic review. Eur Arch Paediatr Dent. 2022 Aug;23(4):501-511. doi: 10.1007/s40368-022-00727-5. Epub 2022 Jul 2. PMID 35779225
- [Background] Keys A, Fidanza F, Karvonen MJ, Kimura N, Taylor HL. Indices of relative weight and obesity. Int J Epidemiol. 2014 Jun;43(3):655-65. doi: 10.1093/ije/dyu058. Epub 2014 Apr 1. PMID 24691951
- [Background] Villa A, Vollemans M, De Moraes A, Sonis S. Concordance of the WHO, RTOG, and CTCAE v4.0 grading scales for the evaluation of oral mucositis associated with chemoradiation therapy for the treatment of oral and oropharyngeal cancers. Support Care Cancer. 2021 Oct;29(10):6061-6068. doi: 10.1007/s00520-021-06177-x. Epub 2021 Mar 31. PMID 33788003
- [Background] Gomaa E, Ayoub MM. Vardenafil oral jellies as a potential approach for management of pediatric irritable bowel syndrome. Saudi Pharm J. 2021 Sep;29(9):955-962. doi: 10.1016/j.jsps.2021.07.020. Epub 2021 Jul 27. PMID 34588841
- [Background] Dastan F, Ameri A, Dodge S, Hamidi Shishvan H, Pirsalehi A, Abbasinazari M. Efficacy and safety of propolis mouthwash in management of radiotherapy induced oral mucositis; A randomized, double blind clinical trial. Rep Pract Oncol Radiother. 2020 Nov-Dec;25(6):969-973. doi: 10.1016/j.rpor.2020.09.012. Epub 2020 Oct 3. PMID 33100913
- [Background] Ibrahim SS, Hassanein FEA, Zaky HW, Gamal H. Clinical and biochemical assessment of the effect of glutamine in management of radiation induced oral mucositis in patients with head and neck cancer: Randomized controlled clinical trial. J Stomatol Oral Maxillofac Surg. 2024 Jun;125(3S):101827. doi: 10.1016/j.jormas.2024.101827. Epub 2024 Mar 15. PMID 38493953
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK565848/